CLINICAL TRIAL: NCT00045617
Title: A Phase II Trial of Patients With Limited Stage Small Cell Lung Cancer Treated With Thoracic Radiation Therapy and Chemotherapy With Cisplatin/Etoposide Followed by Cisplatin/Etoposide and Anti-Idiotype Monoclonal Antibody Vaccines
Brief Title: S0122: Combination Chemotherapy, Radiation Therapy, and Vaccine Therapy in Limited-Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to lack of drug availability.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000256922; S0122 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cisplatin and etoposide followed by vaccine (Experimental): standard chemotherapy with cisplatin and etoposide followed by cisplans and etoposide with an anti-idiotype monoclonal antibody vaccine
  Interventions: Biological: monoclonal antibody 11D10 anti-idiotype vaccine; Biological: monoclonal antibody GD2 anti-idiotype vaccine; Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy

INTERVENTIONS:
Biological: monoclonal antibody 11D10 anti-idiotype vaccine
Biological: monoclonal antibody GD2 anti-idiotype vaccine
Drug: cisplatin
Drug: etoposide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high energy x-rays to damage tumor cells. Vaccines may make the body build an immune response to kill tumor cells. Combining chemotherapy and radiation therapy with vaccine therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining chemotherapy and radiation therapy with vaccine therapy in treating patients who have limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of cisplatin, etoposide, and thoracic radiotherapy followed by cisplatin, etoposide, monoclonal antibody 11D10 anti-idiotype vaccine (TriAb), and monoclonal antibody GD2 anti-idiotype vaccine (TriGem), in terms of overall and progression-free survival of patients with limited stage small cell lung cancer.
* Determine the immune response to each of the 2 anti-idiotype vaccines when used in this regimen in these patients.
* Determine the qualitative and quantitative toxicity of this regimen in these patients.
* Determine the response rates (confirmed and unconfirmed, complete and partial) in patients with measurable disease treated with this regimen.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive cisplatin IV over 1 hour on days 1, 8, 29, and 36 and etoposide IV over 1 hour on days 1-5 and 29-33. Thoracic radiotherapy is administered 5 days a week, beginning on day 1 of chemotherapy, for 5 weeks. Patients then undergo radiotherapy boost for 1.5 weeks.

Patients with stable disease or at least partial response proceed to consolidation therapy.

* Consolidation therapy (begins within 3-5 weeks of the last dose of induction chemotherapy or radiotherapy): Patients receive cisplatin IV over 1 hour on day 1 and etoposide IV over 1 hour on days 1-3 of weeks 11 and 14. Patients also receive monoclonal antibody 11D10 anti-idiotype vaccine (TriAb) and monoclonal antibody GD2 anti-idiotype vaccine (TriGem) intradermally on day 1 of weeks 11, 13, 15, and 17 (4 injections) and then monthly subcutaneously for 2 years. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients who achieve complete response after consolidation chemotherapy undergo cranial radiotherapy 5 days a week for 3 weeks.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed limited stage small cell lung cancer (SCLC)
* Evidence of disease by CT scan of the chest
* Measurable or evaluable disease outside of area of prior surgical resection
* No malignant pericardial or pleural effusions (cytologically positive effusions or exudative effusions not attributable to other etiologies)
* No CNS disease by chest CT scan or MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine no greater than upper limit of normal OR
* Creatinine clearance at least 60 mL/min

Other

* No prior hypersensitivity or contraindication to monoclonal antibody 11D10 anti-idiotype vaccine (TriAb), monoclonal antibody GD2 anti-idiotype vaccine (TriGem), or aluminum hydroxide
* No known sensitivity to rodent proteins (i.e., anti-OKT-3, ONCOSCINT scan)
* No grade 1 or greater symptomatic sensory neuropathy
* No other malignancy except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, adequately treated stage I or II cancer in complete remission, or any other cancer for which patient has been disease free for 5 years
* If significant clinical hearing loss already present, must accept risk of further hearing loss
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for SCLC
* No prior TriAb or TriGem
* No prior murine antibodies
* No prior mouse proteins
* At least 30 days since prior immunotherapy
* At least 30 days since any prior immunization

Chemotherapy

* No prior systemic chemotherapy for SCLC
* No concurrent cyclophosphamide or methotrexate

Endocrine therapy

* At least 30 days since prior systemic corticosteroids
* No concurrent systemic corticosteroids (except as an antiemetic)

Radiotherapy

* No prior radiotherapy to the thorax or neck region
* No concurrent intensity modulated radiotherapy

Surgery

* See Disease Characteristics
* At least 2 weeks since prior thoracic or other major surgery and recovered

Other

* At least 30 days since prior investigational agents or devices
* No other concurrent investigational agents
* No other concurrent immunosuppressants (e.g., cyclosporine)
* No concurrent chronic systemic antihistamines
* No concurrent amifostine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-01; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
overall survival | up to 5 years
  time from date of registration to date of death

SECONDARY OUTCOMES:
immune response | at Week 10
  T-cell proliferation and HAMA testing
toxicity assessment | 22 weeks
  assessment of qualitative and quantitative toxicities
response | 25 weeks
  RECIST partial and complete response

CONTACTS AND LOCATIONS:
Overall Officials: Abdul-Rahman Jazieh, MD, MPH, Study Chair — Barrett Cancer Center
Locations (100):
- United States (99):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Health Science Center, Aurora, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Oregon Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada